CLINICAL TRIAL: NCT04367454
Title: Life-Saving Procedures Performed in the Pre-Decontamination Area While Wearing CBRNe Personal Protective Equipment: A Manikin Randomized Trial
Brief Title: Procedures While Wearing CBRNe Protective Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Matteo Paganini, Principal Investigator, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AOPD 0045954
Record Dates: First submitted 2020-04-22; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Cardiac Arrest; Pneumothorax; Hemorrhage
MeSH Terms: conditions — Heart Arrest; Pneumothorax; Hemorrhage

STUDY DESIGN:
Intervention Model Description: single-center, randomized (1:1), parallel-group, manikin trial
Who Masked: Outcomes Assessor
Masking Description: Blinding of participants and researchers involved in the experiment is not possible. Only the outcome assessor and data analyst (SS) is kept blinded to the allocation of subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personal Protective Equipment (Experimental): Wearing: Tyvek pro-tech® "C" gear (Bonetti, Milano, Italy), a full visor SGE 400 mask (EN 136:98 CL3) connected to an A2B2E2K2-P3 R filter (Spasciani, Milano, Italy), and well-fitting, non-sterile Mapa Ultranitril 480 gloves (Mapa SAS, Colombes, France).
  Interventions: Other: Use of Personal Protective Equipment
- NO-Personal Protective Equipment (No Intervention): only wearing well-fitting, medical examination nitrile gloves.

INTERVENTIONS:
Other: Use of Personal Protective Equipment — As described in the arm descriptions
  Arms: Personal Protective Equipment

SUMMARY:
Out-of-hospital care during Chemical-Biological-Radiological-Nuclear-explosive (CBRNe) events have recently evolved, but the available knowledge is still extremely partial. In particular, the debate is still ongoing regarding which life-saving maneuvers should be implemented in the pre-decontamination phase while wearing CBRNe personal protective equipment (PPE). The investigators hypothesized that PPE may lengthen the execution times and worsen the success rate of invasive and non-invasive procedures.

This trial involves residents in emergency medicine and anesthesia/critical care of the University of Padova (Italy) with the following procedures performed on high-fidelity manikins, after being divided into two groups (wearing and not wearing PPE): positioning of peripheral venous access; intraosseous access; drug preparation and administration; tension pneumothorax (PNX) needle decompression; tourniquet positioning; chest compressions. The primary outcome was the chest compressions depth mean difference between the two groups. As secondary outcomes, the investigators measured differences between the two groups in: the percentages of correct release during chest compressions; chest compressions rate (beats per minute); and the times needed to complete the above-mentioned procedures (other than chest compressions).

The investigators expect that PPE will reduce CPR quality or delay the completion of the procedures.

DETAILED DESCRIPTION:
This is a single-center, randomized (1:1), parallel-group, manikin trial comparing times of execution and quality of life-saving procedures performed by residents while wearing PPE for CBRNe events versus no PPE. The trial was deemed exempt from review by the local Ethics Committee (No. 0045954/2019). The study was conducted aiming to reduce carbon footprint and increase sustainability.

Study Population The trial involves Senior Emergency Medicine (EM) and Anesthesiology and Critical Care (ACC) residents (PGY-4 and -5) from the residency programs of the University of Padova (Padova, Italy), recruited via email by the study coordinator (GM) without selection. Eligible residents are certified as proficient at the procedures described in the next section by the respective residency board, being this a prerequisite to qualify as a PGY-4 and -5 in Italy. The subjects participating in the study don't receive any incentives. Written consent is asked prior to the beginning. The study is organized at the "SIMULARTI" medical simulation center of the University of Padova in Padova, Italy.

Interventions and Procedures Residents are involved in performing the following procedures on the ground on high fidelity manikins: two rescuers CPR (SUSIE - Gaumard Scientific, Miami, FL); tactical tourniquet application (with a Combat Application Tourniquet®, CAT Resources, Rock Hill, SC; on a Trauma Hal - Gaumard Scientific, Miami, FL); tension PNX needle decompression (Truman Trauma X - TruCorp, Lurgan, N. Ireland); positioning of peripheral venous access, intraosseous vascular access (with EZ-IO® - Teleflex, Wayne, PA), and drug preparation and administration (Code Blue III Adult - Gaumard Scientific, Miami, FL). Each procedure is accomplished by the algorithms collected in an operations manual made available to the researchers only, and verbally disclosed to the participants before their attempt (see Online Supplement 1). The participants do not receive any feedback, neither verbal nor visual, during the execution of the procedures. Subjects in the intervention group wear a Tyvek pro-tech® "C" gear (Bonetti, Milano, Italy), a full visor SGE 400 mask (EN 136:98 CL3) connected to an A2B2E2K2-P3 R filter (Spasciani, Milano, Italy), and well-fitting, non-sterile Mapa Ultranitril 480 gloves (Mapa SAS, Colombes, France). Subjects in the control group only wear well-fitting, medical examination nitrile gloves.

After the end of the procedures under investigation, participants from the control group are given the possibility to perform the procedures wearing CBRNe PPE, since this is a training session part of their curricular activities. Finally, an anonymous questionnaire was administered to the participants to evaluate their perception of the experience (Online Supplement 2). The questionnaire was composed of 10 items - 7 positive and 3 negative - that participants had to rate using a 5 point Likert scale (1=totally disagree; 2=disagree; 3=uncertain; 4=agree; 5=totally agree). The internal consistency of the questionnaire was measured using Cronbach's alfa.

Randomization For the 1:1 allocation of the residents, a computer-generated list of random numbers is used. Participants are randomly assigned following variable block sizes of 2 and 4 to either the intervention group (in which they wore CBRNe PPEs) or to a control group (in which they used only one pair of nitrile gloves) (Figure 1). Also, the participants perform each procedure in a random order according to a computer-generated sequence. Randomization is prepared by a researcher not directly involved with the experiments. The allocation of subjects and order of the procedures are concealed by using sequentially numbered, opaque, stapled envelopes, and upheld until each participant was in the simulation rooms. The experiment coordinator (MP) opens the envelopes and assigns participants to group and procedures. Blinding of participants and researchers involved in the experiment is unfortunately not possible. Only the outcome assessor and data analyst (SS) is kept blinded to the allocation.

Outcomes The primary outcome is the difference in sternum to spine chest compressions (CCs) depth during CPR between the two groups. Secondary outcomes are the differences in CCs average rates per minute, percentage of CCs full release, times for completion of tourniquet positioning, PNX decompression, positioning of a peripheral venous catheter and intraosseous access, and drug preparation and administration. As tertiary outcome, the overall participants' perception of this CBRNe simulated training at the end of the session is measured.

Data Collection In each scenario, a researcher collects times with a stopwatch and monitors the correct execution of procedures. In case of errors, the participant is stopped and granted a second attempt, but is excluded from the study. As for CPR, data are collected using UNI® Unified Simulator Control Software ver 2.41.1.0 (Gaumard Scientific, Miami, FL).

Sample Size and Statistical Analysis The investigators calculated that group sample sizes of 18 and 18 would be required to detect a difference of 5.0 mm in CCs depth with a standard deviation (SD) of 5.0 mm, at a significance level (alpha) of 0.05 and at least 80% power, using a two-sided Mann-Whitney test, assuming that the actual distribution could be non-normal. Qualitative data are analyzed descriptively through their distribution frequency. Quantitative data are tested with a Shapiro-Wilk test for normality. Results are presented as mean with SD, and differences tested with independent t-test in case of normally distributed data with equal variance (tested with Levene's test; if not true: Welch test). Otherwise, results are presented as median and interquartile range (IQR), and differences are tested using a Mann-Whitney test. All tests are two-sided and p values <0.05 are considered statistically significant. An estimated difference with 95% confidence interval (CI) is reported for the difference between testing conditions. Statistical software JASP (ver 0.11.1; JASP Team, 2019) is used to analyze the results.

ELIGIBILITY:
Inclusion Criteria:

* Senior Emergency Medicine (EM) and Anesthesiology and Critical Care (ACC) residents (PGY-4 and -5) from the residency programs of the University of Padova (Padova, Italy)

Exclusion Criteria:

* not giving informed consent
* not willing to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
chest compressions | during procedures
  difference in sternum to spine chest compressions depth during CPR

SECONDARY OUTCOMES:
average rates | during procedures
  differences in chest compressions average rates per minute during CPR
chest full release | during procedures
  differences in percentage of chest compressions full release during CPR
tourniquet positioning | during procedures
  differences in times for completion of tourniquet positioning
pneumothorax decompression | during procedures
  differences in times for completion of pneumothorax decompression
venous catheter positioning | during procedures
  differences in times for the positioning of a peripheral venous catheter
intraosseous access positioning | during procedures
  differences in times for the positioning of an intraosseous access
drug preparation and administration | during procedures
  differences in times for drug preparation and administration

OTHER OUTCOMES:
Questionnaire | At the end of the simulations (about 3 hours after the beginning)
  overall participants' perception of the CBRNe simulated training, on a 5 points Likert scale from a minimum of 1 (completely disagree) to a maximum of 5 (completely agree).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Fabris, MD, Study Chair — University of Padova
Locations (1):
- SIMULARTI Simulation Centre, Padua, Veneto, Italy

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year after publication
Access Criteria: Upon request

REFERENCES:
- [Derived] Mormando G, Paganini M, Alexopoulos C, Savino S, Bortoli N, Pomiato D, Graziano A, Navalesi P, Fabris F. Life-Saving Procedures Performed While Wearing CBRNe Personal Protective Equipment: A Mannequin Randomized Trial. Simul Healthc. 2021 Dec 1;16(6):e200-e205. doi: 10.1097/SIH.0000000000000540. PMID 33428358